CLINICAL TRIAL: NCT06893848
Title: Culture Care Program: a Mixed-methods Study Evaluating the Effect of an Innovative In-hospital Experience on Patient Mobility After Thoracic or Abdominal Surgery
Brief Title: Influence of the Culture Care Program on Patient Mobility After Thoracic or Abdominal Surgery: a Mixed-methods Study
Acronym: CULTURECARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haute Ecole ARC Sante (Other)
Responsible Party: Principal Investigator, Dugernier Jonathan, Dr, Haute Ecole ARC Sante
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Study 2024-02620
Record Dates: First submitted 2025-03-07; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Thoracic Surgery; Abdominal Surgery Patients; Hospital Mobility; Mobility Limitation
Keywords: Physical activity; Postoperative recovery; Accelerometer; Early mobilization
MeSH Terms: conditions — Mobility Limitation; Motor Activity

STUDY DESIGN:
Intervention Model Description: The first part of this project is a quantitative monocentric, non-randomized controlled study comparing a group of participants before implementation of the Culture Care program (control group) with a group of participants after implementation of the Culture Care program (Culture Care group). Participants are hospitalized patients and the healthcare workers.
  The second part of this project is a qualitative study once the Culture Care program is implemented.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group of patients (No Intervention): Patients hospitalized after thoracic or abdominal surgery in a conventional in-hospital environment (not modified, before the implementation of the Culture Care program). Patients will receive standard of care, including early mobilization prescribed by the physician according to the ERAS guidelines.
- Culture Care group of patients (Experimental): Patients hospitalized after thoracic or abdominal surgery in an in-hospital environment modernized by the Culture Care program. As with control patients, patients in the Culture Care group will receive the similar standard of care, including early mobilization prescribed by the physician according to the ERAS guidelines.
  Interventions: Other: Culture Care program
- Control group of healthcare workers (No Intervention): Healthcare workers working in the surgical units, with a conventional in-hospital environment (before implementation of the Culture Care program)
- Culture Care group of healthcare workers (Experimental): Healthcare workers working in the surgical units, with an in-hospital environment modernized by the Culture Care program
  Interventions: Other: Culture Care program

INTERVENTIONS:
Other: Culture Care program — The Culture Care program modernizes the in-hospital environment by including art and culture proposed in the form of an individualized pathway. It will be offered primarily to hospitalized patients, but also available to families, caregivers and healthcare professionals. It will aim to create a new hospital experience, different from the one we've always known.
  The Culture Care program will display posters illustrating works of art (paintings, drawings, photographs, etc.) along the hallways. These posters will be interactive, so that a QR code can be scanned to access musical content and audio podcasts (interviews and documentaries) accessible via bone-conduction headphones.
  The Culture Care program is likely to reduce the sedentary behavior of hospitalized patients, by providing an attractive in-hospital environment that is likely to produce both physical and psychological benefits.
  Arms: Culture Care group of healthcare workers; Culture Care group of patients

SUMMARY:
A sedentary behavior in the postoperative phase has a negative impact on recovery from various types of surgery (e.g. abdominal, pulmonary, cardiac or esophageal). In fact, sedentary behavior in the days following surgery is associated with an increased risk of postoperative complications, longer hospital stays and, consequently, higher healthcare costs. Stimulating early mobilization and increasing the level of physical activity after surgery therefore remains a relevant current challenge. The Culture Care program will propose a new experience of the hospital towards an attractive and stimulating intrahospital environment, including art and culture. The hypothesis is that the innovative, positive hospital experience offered by the Culture Care program could contribute to increasing patients' mobility in the postoperative phase and thus reduce the sedentary behaviour compared with a control group included before the implementation of the program.

The aim of this study is to explore the effect of the Culture Care program (Control group versus Culture Care group) on the mobility of patients hospitalized after thoracic or abdominal surgery, by determining the level of prediction in relation to the influencing covariates reported in the literature.

The first quantitative part of this research project will compare the mobility of patients hospitalized after surgery, before (control group) and after the implementation of the Culture Care program (Culture Care group). Patients will be asked to wear an accelerometer for the first five post-operative days, and to complete three questionnaires (psychological well-being, physical recovery, perception of their mobility).

Healthcare workers will be asked to complete a survey on their readiness to stimulate patients' mobility before and after the Culture Care program.

The second part will be qualitative including individual semi-structured interviews with patients and healthcare workers during the Culture Care program, to gather their experiences.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Surgical Units in the Surgical Department of the Hôpital de Neuchâtel implementing the Culture Care program.
* Elective thoracic or abdominal surgery with an expected hospital stay of at least 2 days (i.e. discharge on postoperative day 3).
* Neurocognitive and physical ability to complete questionnaires and individual participation in the Culture Care program.
* Full capacity of discernment and signed informed consent to participate in the study.

Exclusion Criteria:

* Outpatient surgery.
* Emergency surgery.
* Mobility severely impaired prior to surgery: patients with 1 or 2 lower-limb amputations, patients with wheelchair mobility only, neurodegenerative diseases.
* Bed restiction between POD 1 and POD 5 for medical reasons, i.e. surgery, post-operative complications or other pre-existing cardiorespiratory, neurological or orthopedic reasons.
* Transfer to ICU
* Only during the Culture Care phase, an unplanned transfer to another unit that does not have the Culture Care program (e.g. Medicine units).
* Technical problem with the accelerometer (e.g. disfunctioning battery).
* Allergic reaction to any dressing used to attach the accelerometer.
* End-of-life patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Daily time spent out of bed | From postoperative day 1 to postoperative day 3.
  This outcome will be assessed by accelerometry
Daily steps number | From postoperative day 1 to postoperative day 3.
  This outcome will be assessed by accelerometry

SECONDARY OUTCOMES:
Number of patients mobilized on the day of surgery | The day of surgery (Day 0)
  Out of bed: sitting in the chair, standing, walking, etc. This outcome will be assessed by accelerometry.
Daily steps number | From postoperative day 1 to postoperative day 5.
Mean daily duration of physical inactivity, light physical activity and moderate-to-vigorous physical activity | From postoperative day 1 to postoperative day 5.
Quality of recovery after surgery | At postoperative day 2 and at discharge (maximum 1 day before)
  This outcome will be assessed using the Quality of Recovery in 15 questions questionnaire (QoR-15) with a 11-point numerical rating scale with a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery)
Psychological well-being | At postoperative day 2
  This outcome will be assessed using the Hospital Anxiety and Depression scale to measure anxiety and depression, with a score of 0 to 7 considered normal, 8 to 10 indicate mild symptoms, 11 to 14 indicate moderate symptoms and 15 to 21 indicate severe symptoms.
Experience of in-hospital mobility | At postoperative day 2
  This outcome will be assessed using a survey with Likert scale questions with seven point scale to express how much they agree or disagree with different statements about barriers and facilitators to mobility during the hospital stay.
  In addition, patients will be asked to rate their satisfaction about the in-hospital environment (with 0 being the lowest and 10 being the highest).
Postoperative complications rate | From the day of surgery to hospital discharge (from maximum 1 day before discharge to 2 days after discharge)
  This outcome will be assessed using the Comprehensive Complications Index (CCI®), a score ranging from 0 (no complication) to 100 (death).
Length of hospital stay | At hospital discharge (from maximum 1 day before discharge to 2 days after discharge)
Number of patients with adverse events | At hospital discharge (from maximum 1 day before discharge to 2 days after discharge)
  Adverse events related to early mobilization of patients in the postoperative phase up to discharge, i.e. number of falls or loss of consciousness, accidental removal of drains or catheters
Number of adverse events per patients | At hospital discharge (from maximum 1 day before discharge to 2 days after discharge)
  Adverse events related to early mobilization of patients in the postoperative phase up to discharge, i.e. number of falls or loss of consciousness, accidental removal of drains or catheters
Perception of the work environment and readiness to stimulate the mobility of hospitalized patients after surgery | During the 2 month period before the implementation of the Culture Care. This outcome will be assessed 3 month after the implementation of the Culture Care program.
  This outcome will be assessed among the healthcare workers via a survey.

OTHER OUTCOMES:
Patients experience of the Culture Care intervention | Interviews will start after the end of the quantitative study, for a anticipated duration from 1 to 5 months, maximum 8 months). Interviews will be conducted with patients between postoperative day 2 and postoperative day 5.
  Semi-structured interview (for the intervention group)
Healthcare workers experience of the Culture Care intervention | Interviews will start after the end of the quantitative study, for an anticipated duration from 1 to 5 months, maximum 8 months)
  Semi-structured interview (for the intervention group only) conducted with the healthcare workers working in the units modernized with the Culture Care program.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de Neuchâtel, Neuchâtel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided